CLINICAL TRIAL: NCT05412524
Title: Impact of Reading on Endogenous Oxytocin System of Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kelsey Sullivan, MD, 4th Year Resident, Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR220058
Record Dates: First submitted 2022-05-10; First posted 2022-06-09 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Premature Infant Disease; Development, Infant

STUDY DESIGN:
Intervention Model Description: Mothers and, if desired, mother's partner will read to preterm infant as frequently and as much as they are able to. Reading is the intervention. The variable of interest is parents' and infants' change in salivary oxytocin receptor gene methylation (OXTRm) over time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reading (Experimental): Mother and, if desired, mother's partner will read to infant for at least 15 minutes per week, but will be encouraged to read to infant as much as possible. Saliva will be collected from infants and parents for OXTRm assay at pre-specified time points, and at these time point parents will also complete standardized questionnaires including PSS-NICU, PROMIS depression, and PROMIS anxiety to assess parental mood and stress. Reading time will be measured with a reading log provided to the parents, as well as with a commercially-available LENA device to measure word count.
  Interventions: Behavioral: reading

INTERVENTIONS:
Behavioral: reading — Mothers and, if desired, mother's partner will read to preterm infant as frequently and as much as they are able to. Reading is the intervention. The variable of interest is parents' and infants' change in salivary oxytocin receptor gene methylation (OXTRm) over time.

SUMMARY:
The purpose of this study is to learn how early language exposure may be related to changes in DNA in parents and their premature infants. While a person's genetic code is determined at the time of conception, the way that some genes are expressed in the body can be changed even after an individual is born. These changes are called epigenetic changes. In this study, the investigators want to learn about the epigenetic changes that happen after a premature baby is born and whether a parent's interaction with their baby can influence these epigenetic changes. The investigators will look at epigenetic changes by collecting saliva samples from parents and their preterm babies, here defined as babies born at <33 weeks gestation. Specifically, the investigators will be looking at salivary levels of DNA methylation of the oxytocin receptor gene (OXTRm). The investigators will track changes in OXTRm levels over time in parents and their babies and see if these levels change in relation to how much time parents spend with their babies and how much time they spend reading to their babies. The investigators will ask mothers and, if desired, their partners to read to their babies for at least 15 minutes per week. The investigators will ask them to track time spent with the baby and reading time on a log, and will also measure word count with a commercially-available LENA device. The investigators will use logistic regression analysis to identify the independent association between OXTR DNA methylation and time spent with parent(s) and word count.

DETAILED DESCRIPTION:
Student's t-test and Pearson's chi-square tests will be used to compare continuous and categorical variables, respectively. Logistic regression analysis will used to identify the independent association between OXTR DNA methylation and time spent with parent(s) and word count. Variables with p≤0.20 in the univariate analysis will be entered into a stepwise logistic multivariate regression model. Odds ratios with 95% confidence intervals will be calculated. p value of less than 0.05 will be considered statistically significant.

A protocol modification was submitted to and approved by the University of Virginia IRB due to slower than expected participant enrollment. The protocol was modified such that:

* Enrollment of <33 week instead of <32 week infants was permitted
* Enrollment was permitted through the first 2 weeks after birth instead of through the first 1 week after birth

ELIGIBILITY:
Inclusion Criteria:

* Infants <33 week gestational age at birth
* Mother must be able to visit at least once per week
* Mother or primary caregiver must participate; father or secondary caregiver may participate as well
* Mother must commit to minimum of 15 minutes reading at least once per week

Exclusion Criteria:

* Infant with life-limiting conditions
* Mother is non-English speaking
* Illiteracy of mother

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Salivary oxytocin receptor gene DNA methylation (OXTRm) | Birth to discharge from neonatal intensive care unit (approximately 1-4 months)
  Salivary oxytocin receptor gene DNA methylation (OXTRm), change in time as related to amount of time parents spend reading to infant

SECONDARY OUTCOMES:
Parental stress | Birth to discharge from neonatal intensive care unit (approximately 1-4 months)
  Parental stress, as measured by PSS-NICU, and its correlation with amount of time parents spend reading to infants
Parental depression | Birth to discharge from neonatal intensive care unit (approximately 1-4 months)
  Parental stress, as measured by the PROMIS depression short form, and its correlation with amount of time parents spend reading to infants
Parental anxiety | Birth to discharge from neonatal intensive care unit (approximately 1-4 months)
  Parental stress, as measured by the PROMIS anxiety scale, and its correlation with amount of time parents spend reading to infants

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perkeybile AM, Carter CS, Wroblewski KL, Puglia MH, Kenkel WM, Lillard TS, Karaoli T, Gregory SG, Mohammadi N, Epstein L, Bales KL, Connelly JJ. Early nurture epigenetically tunes the oxytocin receptor. Psychoneuroendocrinology. 2019 Jan;99:128-136. doi: 10.1016/j.psyneuen.2018.08.037. Epub 2018 Aug 31. PMID 30227351
- [Background] Caskey M, Stephens B, Tucker R, Vohr B. Adult talk in the NICU with preterm infants and developmental outcomes. Pediatrics. 2014 Mar;133(3):e578-84. doi: 10.1542/peds.2013-0104. Epub 2014 Feb 10. PMID 24515512
- [Background] Krol KM, Moulder RG, Lillard TS, Grossmann T, Connelly JJ. Epigenetic dynamics in infancy and the impact of maternal engagement. Sci Adv. 2019 Oct 16;5(10):eaay0680. doi: 10.1126/sciadv.aay0680. eCollection 2019 Oct. PMID 31663028
- [Background] Caskey M, Stephens B, Tucker R, Vohr B. Importance of parent talk on the development of preterm infant vocalizations. Pediatrics. 2011 Nov;128(5):910-6. doi: 10.1542/peds.2011-0609. Epub 2011 Oct 17. PMID 22007020
- [Background] Neri E, De Pascalis L, Agostini F, Genova F, Biasini A, Stella M, Trombini E. Parental Book-Reading to Preterm Born Infants in NICU: The Effects on Language Development in the First Two Years. Int J Environ Res Public Health. 2021 Oct 29;18(21):11361. doi: 10.3390/ijerph182111361. PMID 34769878